CLINICAL TRIAL: NCT06346457
Title: The Impact of Anti-estrogenic Therapy in Breast Cancer Patients on Brain Architecture, Psychosexual Health, and Quality of Life
Brief Title: Breast Cancer & Antiestrogenic Therapy & Brain
Status: Not yet recruiting | Type: Observational
Sponsor: International Research Training Group 2804 (Other)
Collaborators: German Research Foundation (Other); University Hospital Tuebingen (Other); Uppsala University (Other)
Responsible Party: Sponsor
Other Study IDs: IRTG_P08
Record Dates: First submitted 2024-02-14; First posted 2024-04-04 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-03

CONDITIONS: Breast Cancer Female; Healthy Female; Menopause; Anti-estrogenic Therapy
Keywords: Women´s mental health; Breast cancer; Anti-estrogenic therapy; Neuroimaging(fMRI); Estrogen; Menopause; Reward processing; Psychosexual health; Quality of life (QoL); MRI
MeSH Terms: conditions — Breast Neoplasms | interventions — Tamoxifen; Letrozole; Gonadotropin-Releasing Hormone

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- premenopausal women diagnosed with breast cancer: receiving anti-estrogenic therapy
  Interventions: Drug: Tamoxifen
- postmenopausal women diagnosed with breast cancer, with/out previous hormonal replacement therapy: receiving anti-estrogenic therapy
  Interventions: Drug: Letrozole; Drug: Letrozole + GnRH
- premenopausal healthy women: before menopause
- postmenopausal healthy women with/out previous hormonal replacement therapy: after menopause

INTERVENTIONS:
Drug: Tamoxifen — Tamoxifen is 20 mg once daily for two to three weeks.
  Groups: premenopausal women diagnosed with breast cancer
Drug: Letrozole — Letrozole (Aromatase inhibitor) is 2,5 mg once daily for two to three weeks.
  Groups: postmenopausal women diagnosed with breast cancer, with/out previous hormonal replacement therapy
Drug: Letrozole + GnRH — When they take Letrozole + GnRh, the GnRh is an injection once a month.
  Groups: postmenopausal women diagnosed with breast cancer, with/out previous hormonal replacement therapy

SUMMARY:
The study aims to investigate the effect of anti-estrogenic therapy in breast cancer patients on neural reward processing, psychosexual health, and quality of life, in reproductive vs. menopausal women. The investigators are directly comparing four groups 1) premenopausal women diagnosed with breast cancer receiving anti-estrogenic therapy, 2) postmenopausal women diagnosed with breast cancer with and without previous hormonal replacement therapy, receiving anti-estrogenic therapy, 3) premenopausal healthy women, and 4) postmenopausal healthy women. Furthermore, via assessment and integration of various data including subjective/self-report data via questionnaires and a standardized interview, physiological/endocrine (via blood sample), psychological and neural data (including anatomical scans, Diffusion tensor imaging (DTI), resting state, and a reward processing paradigm), this project will shed light on the connection between the brain, anti-estrogenic therapy, and psychosexual health.

DETAILED DESCRIPTION:
If participants qualify for the current study, the investigators will invite them to the laboratory (T0), where participants will provide written, informed consent. Subsequently, the investigators will conduct a standardized clinical interview to screen for mental disorders (SCID-5-CV). Participants will also be informed about the study procedure. After the interview, participants will receive a password-protected link by email to access an online survey that measures, among other things, depressive symptoms, personality traits, gender identity and norms, relationship quality, sexual health, state and trait anxiety, and verbal intelligence.

All fMRI measurements (T1 and T2) will precede the hormonal and surgical components of the breast cancer treatment. Biopsy and analysis of tumor tissue will be performed in the pathology department of the University of Tuebingen Women's Clinic. Similarly, clinical routine procedures and adjuvant systemic treatment will be administered at the University of Tuebingen Women's Clinic.

Following the first interview, participants will undergo the first MRI session (T1) before starting anti-estrogenic therapy. The second MRI session (T2) will be scheduled two- three weeks after commencing anti-estrogenic therapy and before the surgery.

For controls, premenopausal women and postmenopausal women who have stopped or never used hormone replacement therapy will be included. At the start of the MRI sessions, a 30ml blood draw will be performed by medically trained personnel. The investigators anticipate hormonal changes between T1 and T2 due to breast cancer treatment (anti-estrogenic therapy).

After the second measurement (T2), women diagnosed with breast cancer will be invited to the third online session (T3) to assess possible related changes in psychosexual health, body image, and quality of life through questionnaires.

The investigators have meticulously planned the sequence of our MRI measurements to ensure a comprehensive exploration of various aspects of brain structure and function. The protocol is structured as follows:

1. Anatomical Scan: The session begins with an anatomical scan, aiming to provide detailed insights into the structural aspects of the brain. This foundational step allows for a precise understanding of the anatomical features before delving into functional assessments.
2. Resting State: Following the anatomical scan, participants will engage in a resting-state session lasting approximately 10 minutes. During this period, participants will watch a video to capture diverse facets of brain function and physiological states during rest. Resting-state measurements provide valuable information about intrinsic brain activity in the absence of a specific task.
3. Effort Allocation Task (EAT): Subsequent to the resting-state session, participants will undertake the effort allocation task (EAT). This task is strategically designed to explore the trade-off between the benefits of effort and the associated costs. Participants will be involved in a task where monetary points are at stake, requiring physical effort by manipulating a grip-force measuring device. The payoff will be proportional to the duration of their invested effort. The EAT is anticipated to last up to 17 minutes.
4. Diffusion Tensor Imaging (DTI): Following the EAT, participants will undergo Diffusion Tensor Imaging (DTI) to examine and map the white matter tracts in the brain. DTI is a sophisticated imaging technique that provides insights into the microstructural organization of white matter pathways, offering valuable information about connectivity.

This sequential approach from anatomical scanning to resting state, effort allocation task, and DTI is designed to systematically investigate both the structural and functional aspects of the brain in our study participants. The combination of these different imaging modalities enables a comprehensive understanding of the neural dynamics associated with anatomical structures, intrinsic brain activity at rest, responses to effortful tasks, and the organization of white matter tracts.

To comprehensively investigate self-report changes, the investigators will administer several questionnaires designed to assess various aspects. These questionnaires will focus on body image, psychosexual health, cancer-related quality of life changes, dyadic adjustment scale, well-being, and positive and negative affect changes. The data will be collected and managed through Redcap, providing a systematic and secure platform for organizing and analyzing participant responses. This approach ensures a thorough exploration of subjective experiences and enables a nuanced understanding of the psychological and emotional impact of the variables under investigation.

To thoroughly investigate cognitive changes, the investigators will use a home-testing battery. Participants will perform two online tasks: a reinforcement-learning risk sensitivity task and a gamified Pavlovian go/no-go task with varied bandits. Both tasks will be conducted weekly for three weeks, totaling approximately 1 hour. Data will be stored at the Quantitative Biology Center (QBiC) at the University of Tuebingen.

ELIGIBILITY:
Inclusion Criteria:

* Women before or after menopause
* With/without a diagnosis of breast cancer
* Between 18 and 70 years old
* Body mass index 18-35 kg/m²
* Fluent in written and spoken German
* At least an intermediate school leaving certificate

Exclusion Criteria:

* Any neurological or mental disease based on standardized diagnoses confirmed via the structured clinical interview for DSM-5, Clinical Version (SCID-5-CV)
* Women who gave birth or were breastfeeding within the last year
* Participants with a history of sexual trauma or abuse
* Participants taking any medication interfering with brain activation
* Participants taking oral contraceptives
* Male breast cancer patients
* Patients with alcohol or substance abuse
* Patients if the origin of the cancer is not in the breast cells
* Patients have any other physical severe diseases (stroke, diabetes, heart attack, etc.)
* Patients currently ongoing chemotherapy
* Participants who did not consent

Additional exclusion criteria for MRI:

* People with non-removable metal objects on or in the body
* Tattoos (if MRI-incompatible according to expert guidelines)
* Pathological hearing or increased sensitivity to loud noises
* Claustrophobia
* Surgery less than three months ago
* Moderate or severe head injury

Ages: 18 Years to 70 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: The study population (breast cancer patients and healthy control) will mainly consist of residents of Tübingen and surrounding areas.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Correlations between antiestrogen hormone therapy and brain function & structure | Measured twice 2-3 weeks apart; approx. 32 minutes each time
  Possible effects of antiestrogen hormone therapy on brain function (functional activation based on BOLD effect) and structure in pre- and postmenopausal women diagnosed with breast cancer. Anatomical scan, Resting state and Diffusion Tensor Imaging will be assessed
Correlations between antiestrogen hormone therapy and reward processing in both behavioral and neural aspects | Measured twice 2-3 weeks apart; approx. 17 minutes each time
  Possible effects of antiestrogen hormone therapy on reward processing in pre- and postmenopausal women diagnosed with breast cancer. Effort Allocation Task will be applied.
Brain Disparities: Contrasting Breast Cancer Patients with Healthy Controls | Measured twice 2-3 weeks apart; approx. 32 minutes each time
  Any differences in brain Function (functional activation based on BOLD effect) between Breast Cancer Patients and Healthy control
Reward Processing Disparities: Contrasting Breast Cancer Patients with Healthy Controls | Measured twice 2-3 weeks apart; approx. 17 minutes each time
  Differences in reward processing between Breast Cancer Patients and Healthy control. Effort Allocation Task will be applied.
Brain Disparities: Contrasting Breast Cancer Patients with Healthy Controls | Measured twice 2-3 weeks apart; approx. 32 minutes each time, with fMRI, Anatomical Scan and Diffusion tensor imagingDiffisuin
  Any differences in brain structure between Breast Cancer Patients and Healthy control.

SECONDARY OUTCOMES:
Correlation between antiestrogen hormone therapy and psychosexual health | Measured three times: before treatment, within 2-3 weeks after treatment and 6 months after treatment; approx 60 minutes each time
  Possible effects of antiestrogen hormone therapy on psychosexual health in pre- and postmenopausal women diagnosed with breast cancer.
  Questionnaires: Body Image Scale, Female Sexual Function Index
Correlation between antiestrogen hormone therapy and quality of life | Measured with questionnaires three times: before treatment, within 2-3 weeks after treatment and 6 months after treatment; approx 60 minutes each time
  Possible effects of antiestrogen hormone therapy on quality of life in pre- and postmenopausal women diagnosed with breast cancer.
  Questionnaires:European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire, Positive and Negative Affect Schedule
Psychosexual Health Disparities: Contrasting Breast Cancer Patients with Healthy Controls | Measured two times: before treatment and within 2-3 weeks after treatment; approx 60 minutes each time
  Differences in Psychosexual health between Breast Cancer Patients and Healthy control.
  Questionnaires: Female Sexual Function Index
Psychosexual Health Disparities: Contrasting Breast Cancer Patients with Healthy Controls | Measured two times: before treatment and within 2-3 weeks after treatment; approx 60 minutes each time
  Differences in Psychosexual health between Breast Cancer Patients and Healthy control.
  Questionnaires: Body Image Scale
Correlation between antiestrogen hormone therapy and cognitive changes | Measured for 2-3 weeks: Patients performing both tasks for 2-3 weeks.
  Possible effects of antiestrogen hormone therapy on cognitive changes in pre- and postmenopausal women diagnosed with breast cancer. It has two different behavioral tasks measured by home battery testing: a reinforcement-learning risk sensitivity task and a Pavlovian go/no-go task.
Quality of Life Disparities: Contrasting Breast Cancer Patients with Healthy Controls | Measured two times: before treatment, within 2-3 weeks after treatment; approx 60 minutes each time
  Differences in quality of life between Breast Cancer Patients and Healthy control. It measured with questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Birgit Derntl, Prof, Principal Investigator — Department of Psychiatry & Psychotherapy, University of Tuebingen; Sara Brucker, Prof, Principal Investigator — Department of Women's Health University Women's Clinic; Markus Hahn, Prof, Principal Investigator — Department of Women's Health University Women's Clinic; Anna Wikman, Prof, Principal Investigator — Department of Women's and Children's Health, Reproductive Health; Ann Christin Kimmig, Dr, Principal Investigator — Department of Psychiatry & Psychotherapy, University of Tuebingen
Locations (1):
- University of Tuebingen; Department of Psychiatry & Psychotherapy Tuebingen, Tübingen, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: Yes